CLINICAL TRIAL: NCT00933582
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study of Single Doses of JNJ-39439335 Versus Single and Multiple Doses of Naproxen Versus Placebo in the Treatment of Painful Osteoarthritis of the Knee: Focus on Treatment Effects and Methodological Advances
Brief Title: A Clinical Study to Investigate the Effect on Pain Relief of a Single Dose of JNJ-39439335 in Patients With Chronic Osteoarthritis Pain of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Associate Director Early Development
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016420
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Knee Pain; Pain Measurement; Naproxen; Placebo; Treatment Outcome
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: JNJ-39439335; Placebo; Naproxen

SUMMARY:
The purpose of this single-center study is to evaluate the potential analgesic effects of a single oral dose (50 mg) of JNJ-39439335, an investigational drug being developed for the treatment of pain in patients with chronic osteoarthritis pain of the knee. The study will also evaluate the pain treatment response assessments and methods being used in this study. Participants will also take naproxen (500 mg) and placebo (an inactive substance) during the study. Pain assessments after taking JNJ-39439335, naproxen and placebo will be compared.

DETAILED DESCRIPTION:
The purpose of this single-center study is to evaluate the potential analgesic effects of a single oral dose of JNJ-39439335 (50 mg), an investigational drug being developed for the treatment of pain, in patients with chronic osteoarthritis pain of the knee. The study will also evaluate the pain treatment response assessments and methods being used in this study. Naproxen (500 mg) will be used as the active control. The hypothesis of the study is that a single 50 mg oral dose of JNJ-39439335 will be superior to placebo in relieving pain in patients with osteoarthritis knee pain following exercise. Patients will receive JNJ-39439335 , placebo (an inactive substance, like a sugar pill), or naproxen (500 mg) in the clinic on Days 1, 15, and 29, based on the randomly assigned (like flipping a coin) treatment sequence. Patients will stay in the clinic for pain assessments up to 4 hours post-dose. At 6 hours post-dose, patients will be discharged from the clinic. Patients will then take naproxen (500 mg) or matching placebo at 12 hours post-dose and continue taking naproxen (500 mg) or matching placebo every 12 hours for the following 6 days. During the study, starting from the first screening visit, patients will be required to discontinue all pain medication and will be encouraged not to take any rescue medication (quick-relief or fast-acting medications that work immediately to relieve pain), especially during the dosing periods, for up to 6 days after each in-clinic study drug dosing on Day 1, Day 15, and Day 29, respectively. When needed, patients may take paracetamol (500 mg per dose for up to a maximum of 2 grams per day) as rescue medication; however, patients are required not to take any rescue medication starting from 12 hours before through 6 hours after the in-clinic dosing on Day 1, Day 15, and Day 29, respectively. Patients' pain will be evaluated for each of the 3 treatments. Safety assessments, including vital signs, physical exams, electrocardiograms and clinical lab tests will be performed at timepoints throughout the patients' study participation. Patients will receive JNJ-39439335 (50 mg), placebo, or naproxen (500 mg) oral tablets on Days 1, 15, and 29, based on the assigned treatment sequence. At 12 hours postdose, patients in the naproxen treatment arm will start self-administering naproxen (500 mg) twice daily for 6 days while patients in the placebo or the JNJ-39439335 treatment arm will take placebo twice daily for 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic osteoarthritis (OA) pain of the knee (on an average of at least 5 days per week for the 3 months prior to screening)
* Patients whose OA pain worsens with exercise
* Patients who have been taking a non-opioid pain medication for OA knee pain daily with benefit for at least 5 days over the week prior to screening
* Women must be postmenopausal or unable to have children
* Otherwise healthy

Exclusion Criteria:

* Patients with orthopedic and/or prosthetic device in the knee
* have significant pain that is not related to the knee, including significant hip or back pain that in the judgement of the investigator will interfere with pain measures at the knee (Patients with OA in both knees will be allowed into the study)
* Unable to discontinue all formulations of prior pain medications other than paracetamol during the study
* Unable to discontinue paracetamol for 12 hours prior to the clinic visits
* Patients with history of active peptic ulceration, active dyspepsia, gastrointestinal bleeding, Crohn's disease, ulcerative colitis, chronic diarrhea esophageal, and gastric or duodenal ulcer within 3 months prior to screening
* Patients who have had surgery for any chronic pain within 3 months prior to Screening or plans for surgery while in the study
* Patients with history of prior diagnosis of inflammatory arthritis including rheumatoid arthritis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Difference (SPID) for pain following exercise using a 0-10 numerical rating scale | At 4 hours after the in-clinic dosing on Days 1, 15, and 29, respectively

SECONDARY OUTCOMES:
2-hour postdose pain intensity difference (at rest, exercise-induced, and change from pre- to post-exercise) | on Days 1, 15, and 29
4-hour postdose SPID (at rest and change from pre-to-post exercise) | on Days 1, 15, and 29
Change from predose WOMAC (the Western Ontario and McMaster Osteoarthritis Index) | On Days 1, 2, 7, 16, 21, 30, and 35
Change from baseline in current pain numerical rating scale (NRS) | on Days 1, 15, and 29
Change from baseline in patient activity | on Days 1 to 7, 15 to 21, and 29 to 35

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.